CLINICAL TRIAL: NCT03145441
Title: The Impact of Pre-emptive Intraoperative Use of Extracorporeal Cytokine Adsorption During Orthotopic Heart Transplantation
Brief Title: Intraoperative Use of Extracorporeal Cytokine Adsorption During Orthotopic Heart Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SU-AITK/VM-2017/1
Record Dates: First submitted 2017-03-23; First posted 2017-05-09 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Cardiac Transplantation; Cardiopulmonary Bypass

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CytoSorb® (Experimental): The CytoSorb® filter will be installed into the cardiopulmonary bypass circle during cardiac transplantation in this study group (30 patients)
  Interventions: Device: CytoSorb®
- Control (No Intervention): No filter will be installed into the cardiopulmonary bypass circle in this group (30 patients).

INTERVENTIONS:
Device: CytoSorb® — CytoSorb® is a biocompatible, high adsorptive polymer indicated in conditions where cytokine levels are extremely elevated.
  Arms: CytoSorb®

SUMMARY:
There are several factors initiating cytokine storm and dysregulated systemic inflammatory response during cardiac transplantation. This may lead to serious perioperative complications: circulatory collapse, respiratory insufficiency, acute renal and liver failure, multi-organ dysfunction etc.

On the other hand the high level of cytokines may play an important role in the development of graft rejection which is still a relevant problem in this patient group.

There are some new data showing that the use of extracorporeal cytokine adsorber during long cardiopulmonary bypass time (>120min) may be beneficial to prevent SIRS (Systemic Inflammatory Response Syndrome) with decreasing the level of cytokines in patients undergoing elective cardiac surgery. However there is lack of data and studies regarding the effect of extracorporeal cytokine adsorption during cardiac transplantation.

The aim of the study is to investigate the effect of extracorporeal cytokine adsorber built in the cardiopulmonary bypass circle during heart transplantation. The hypothesis is that removal of cytokines during heart transplantation prevents the development of extreme systemic inflammatory response, hemodynamic collapse dominated by vasoplegia, and contribute to reduce the incidence of severe perioperative complications and early graft rejection.

DETAILED DESCRIPTION:
Patients undergoing cardiac transplantation will be enrolled in the study after giving a written, signed informed consent.

The participants will be randomized into two groups:

* intervention group (30 patients): a cytokine adsorber (CytoSorb®) will be installed into the cardiopulmonary bypass circle during the operation
* control group (30 patients): no cytokine adsorber will be used during cardiopulmonary bypass

The investigators will collect demographic, clinical and laboratory data about patients before, during and after the operation.

The the use of vasopressors and inotropes in the perioperative period, length of mechanical ventilation, ICU and hospital stay, and incidence of perioperative complications, early cellular or humoral graft rejection, and survival will be documented.

The level of cytokines (IL-1, IL-6, IL-10, IL-17, tumor necrosis factor-alfa) and complements before, during and after the use of cardiopulmonary bypass will be determined if the investigators find relevant difference between the two groups in clinical variables.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing heart transplantation
* no medical or mechanical circulatory support straight before transplantation
* age > 18 years

Exclusion Criteria:

* age < 18 years
* septic condition (controlled infection) before transplantation
* prolonged hospital stay straight before transplantation
* use of positive inotropes or vasopressors straight before transplantation
* use of mechanical circulatory support straight before transplantation
* acute liver or kidney failure straight before transplantation
* high urgency transplantation
* retransplantation
* the patient declines participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Early postoperative hemodynamic instability | 24-48 hours
  Hemodynamic instability described by Vasoactive Inotropic Score and calculated for the first two postoperative days.
  Vasoactive Inotropic Score is considered as 'high' if values ≥ 30 points, representing higher risk for worse outcomes.
Postoperative vasoplegia syndrome | 24-48 hours
  Severity of postoperative vasoplegia based on criteria of vasoplegia syndrome: Norepinephrine reqirements ≥ 0.3 μg/kg/min AND arginine vasopressin requirements at any dose
Cytokine and complement levels | 24-48 hours
  Level of pro- and anti-inflammatory cytokines (IL-1, IL-6, IL-10, IL-17, tumor necrosis factor-alfa) and complements immediately after induction of anesthesia, before initiation of cardiopulmonary bypass (CPB), 2 hours after initiation of CPB, at termination of CPB, 6-12-24 hours after initiation of CPB

SECONDARY OUTCOMES:
Inflammatory reaction | 24-48 hours
  Level of C reactive protein (CRP), white blood cells and procalcitonin immediately after induction of anesthesia, before initiation of cardiopulmonary bypass (CPB), 2 hours after initiation of CPB, at termination of CPB, 6-12-24 hours after initiation of CPB
Mechanical ventilation | up to 6 months
  Length of mechanical ventilation
Hospital stay | up to 6 months
  Length of ICU and hospital stay
Length of survival | 1 year
  Length of survival after heart transplantation
Medical circulatory support | 72 hours
  Use and dosage of vasopressors and inotropes immediately after induction of anesthesia, before initiation of cardiopulmonary bypass (CPB), 2 hours after initiation of CPB, at termination of CPB, 6-12-24 hours after initiation of CPB, on 2nd and 3rd postoperative day
Perioperative complications | up to 1 month
  Incidence of perioperative complications after heart transplantation during ICU stay (sepsis, SIRS, respiratory failure, acute renal failure, acute liver failure, postoperative cognitive dysfunction, graft failure)
The incidence of early rejection | 1 month
  The incidence of early (< 1 month) cellular or humoral rejection after heart transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernardi MH, Rinoesl H, Dragosits K, Ristl R, Hoffelner F, Opfermann P, Lamm C, Preissing F, Wiedemann D, Hiesmayr MJ, Spittler A. Effect of hemoadsorption during cardiopulmonary bypass surgery - a blinded, randomized, controlled pilot study using a novel adsorbent. Crit Care. 2016 Apr 9;20:96. doi: 10.1186/s13054-016-1270-0. PMID 27059056
- [Background] Kellum JA, Venkataraman R, Powner D, Elder M, Hergenroeder G, Carter M. Feasibility study of cytokine removal by hemoadsorption in brain-dead humans. Crit Care Med. 2008 Jan;36(1):268-72. doi: 10.1097/01.CCM.0000291646.34815.BB. PMID 18090355
- [Background] Liang TB, Yu ZY, Zheng SS. [Expression of non-T cell derived cytokines in acute rejection after heart transplantation: experiment with mouse model]. Zhonghua Yi Xue Za Zhi. 2006 Jan 3;86(1):26-30. Chinese. PMID 16606531